CLINICAL TRIAL: NCT03217487
Title: A Randomized Controlled Clinical Trial of Corneal Epithelial Autograft for the Treatment of Limbal Stem Cell Deficiency
Brief Title: Corneal Epithelial Autograft for LSCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chunxiao Wang (Other)
Responsible Party: Sponsor-Investigator, Chunxiao Wang, Clinical investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017KYPJ051
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal epithelial autograft (Experimental): Femtosecond laser assisted corneal epithelial autograft from the other eye in the treatment of LSCD
  Interventions: Procedure: Corneal epithelial autograft; Device: Femtosecond laser
- Limbal conjunctival autograft (Active Comparator): Diamond knife assisted limbal conjunctival autograft from the other eye in the treatment of LSCD
  Interventions: Procedure: Limbal conjunctival autograft; Device: Diamond knife

INTERVENTIONS:
Procedure: Corneal epithelial autograft — Epithelial tissue, equal in area to the diseased eye's cornea bed, will be obtained from the fellow eye using femtosecond laser technology. This corneal epithelial autograft is then ready for transplantation on the disease eye, following removal of scarred and diseased epithelium.
  Arms: Corneal epithelial autograft
Procedure: Limbal conjunctival autograft — A 3- to 5- clock hour limbal-conjunctival autograft will be obtained from the fellow eye. This is then ready for transplantation on the disease eye following removal of scarred and diseased epithelium.
  Arms: Limbal conjunctival autograft
Device: Femtosecond laser — A commercial femtosecond laser to create a particular shaped graft for transplantation
  Arms: Corneal epithelial autograft
Device: Diamond knife — A diamond knife to create a particular shaped limbal graft for transplantation
  Arms: Limbal conjunctival autograft

SUMMARY:
The purpose of the study is to explore whether femtosecond laser-assisted corneal epithelial autograft is more effective than limbal conjunctival autograft for ocular surface reconstruction in patients with limbal stem cell deficiency (LSCD).

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral LSCD secondary to ocular burns, with the duration of disease of at least 24 months at the time of screening visit;
2. Presence of superficial neo-vascularization affecting at least 2 cornea quadrants and involving central cornea;
3. Informed consent signed by patient or legal guardian. Having the ability to comply with study assessments for the full duration of the study.

Exclusion Criteria:

1. LSCD of mild degree, with less than 2 quadrants of neo-vessel invasion and without central cornea involvement;
2. LSCD by ocular surface disorders other than pterygium;
3. Eyelids malposition;
4. The center corneal thickness<450µm, the depth of corneal opacity > 150µm;
5. High myopia with a spherical equivalent of -15.0 D or less;
6. Corneal or ocular surface infection within 30 days prior to study entry;
7. Ocular surface malignancy;
8. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%;
9. Renal failure with creatinine clearance< 25ml/min;
10. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L;
11. Platelet levels < 150,000 or > 450,000 per microliter;
12. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
13. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy;
14. Pregnancy (positive test) or lactation;
15. Participation in another simultaneous medical investigation or clinical trial;
16. Severe cicatricial eye disease; Conjunctival scarring with fornix shortening;
17. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases;
18. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye;
19. Any medical or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent;
20. Signs of current infection, including fever and treatment with antibiotics;
21. Active immunological diseases;
22. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Restoration of corneal surface in the diseased eye | 1 year
  Restoration of a completely epithelized, stable, and avascular corneal surface in the diseased eye.
Restoration of corneal surface in the fellow eye | 1 year
  Restoration of a completely epithelized, stable, and avascular corneal surface in the fellow eye.

SECONDARY OUTCOMES:
Uncorrected and best-corrected visual acuity in both eyes | 1 year
  To measure changes of uncorrected and best-corrected visual acuity using ETDRS chart.
Corneal power, astigmatism and aberration in both eyes | 1 year
  To changes of corneal power, astigmatism and aberration using autorefractor keratometer and wavefront aberrometer respectively.
Corneal sensation in both eyes | 1 year
  To assess corneal sensation using Cochet-Bonnet esthesiometer.
Corneal thickness in both eyes | 1 year
  To measure corneal thickness using anterior segment optical coherence tomography (AS-OCT).
Density of stromal nerve and stromal keratocytes in both eyes | 1 year
  To assessing density of stromal nerve and stromal keratocytes using in vivo confocal microscopy.
Reconstruction of limbal palisades of Vogt in the diseased eye | 1 year
  To assessing reconstruction of limbal palisades of Vogt using in vivo confocal microscopy.
Corneal haze in both eyes | 1 year
  To measuring corneal haze using in vivo confocal microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Ting Huang, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guanzhou, Guangdong, China